CLINICAL TRIAL: NCT01294176
Title: Lipoic Acid as a Treatment for Acute Optic Neuritis: A Pilot Study
Brief Title: Lipoic Acid as a Treatment for Acute Optic Neuritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Vijayshree Yadav, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OHSU IRB00005634
Record Dates: First submitted 2010-08-10; First posted 2011-02-11 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Optic Neuritis
Keywords: Optic Neuritis; Lipoic Acid; Multiple Sclerosis; Antioxidant; OCT; Acute
MeSH Terms: conditions — Optic Neuritis; Multiple Sclerosis | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Lipoic Acid (Active Comparator): Lipoic acid is a natural antioxidant available as an oral dietary supplement. A higher than average dose of 1200mg will be administered in this trial.
  Interventions: Drug: Lipoic Acid
- Avicel™ (Placebo Comparator): The placebo is Avicel™ (microcellulose crystal) and 4.3 mg quercetin (a bioflavanoid).
  Interventions: Drug: Lipoic Acid

INTERVENTIONS:
Drug: Lipoic Acid — Lipoic acid will be administered orally, in two 600mg capsules, for a total 1200mg dose. The dose will be administered daily for a 6-week treatment period.

SUMMARY:
The purpose of this study is to determine if oral lipoic acid can safely help relieve permanent optic nerve injury in patients diagnosed with acute optic neuritis. It will also explore how the body absorbs and breaks down the study drug, and what effects it has on the immune system.

DETAILED DESCRIPTION:
Oral lipoic acid is an antioxidant that helps proteins work in the body. It is available in oral and intravenous formulations and has been used in the past to treat nerve damage like that seen in diabetes and some other metabolic disorders. It is available as a dietary supplement in the United States.

Patients with a diagnosis of acute optic neuritis who are enrolled in the study will undergo medical and nervous system examinations, and blood draws. The study doctor will take a medical history and perform physical examinations. Research assistants at the MS Center, who are trained in blood draws, will perform the blood draws. Patients will also undergo Optical coherence tomography (OCT) examination at Casey Eye Institute, and receive two MRIs at Oregon Health and Science University (OHSU). Because it is a placebo-controlled trial, subjects will have a 50:50 chance of receiving either placebo (inactive) or study drug. If enrolled in the study, patients will take two gel capsules of the study drug or placebo at the same time every day for six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute, unilateral AON with visual symptoms (vision loss) of 14 days or less
* 18 - 65 years of age, inclusive
* AON as a first event (possibly idiopathic) or in relationship to clinically isolated syndrome or to MS according to McDonald criteria
* No previous history of optic neuritis or ophthalmoscopic signs of optic atrophy in the affected eye
* Subject is available for treatment initiation within 14 days of onset of AON symptoms

Exclusion Criteria:

* Other causes of visual loss in the affected eye (e.g. amblyopia or glaucoma
* OCT is non-evaluable at screening visit due to edema.
* AON symptoms improve before administration of study medication.
* Subject has fever or active infection at time of enrollment.
* Subject is pregnant or breast-feeding.
* Subject has diabetes mellitus.
* Subject has another significant health problem (e.g. active coronary heart disease, liver disease, significant pulmonary disease).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the difference from baseline in retinal nerve fiber layer (RNFL) thickness of the affected optic nerve, as determined by OCT, at 12 and 24weeks post LA treatment. | Baseline, Week 24
  Individual data will be assessed at the last study visit (six months post baseline). Group data cannot be assessed until all participants have exited the study. The time frame for final assessment of the primary outcome measure is dependent on how quickly the recruitment goal is met.

SECONDARY OUTCOMES:
Secondary outcome measures to assess optic nerve injury will be changes from baseline in the RNFL thickness at week 24, and changes from baseline in low- and high-contrast visual acuity, contrast sensitivity, and visual field changes at weeks 12 and 24. | Baseline, Week 24
  Individual data will be assessed at the last study visit (six months post baseline). Group data cannot be assessed until all participants have exited the study. The time frame for final assessment of the primary outcome measure is dependent on how quickly the recruitment goal is met.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States